CLINICAL TRIAL: NCT02279550
Title: Institutional Registry of Hip Fracture in the Elderly
Status: Recruiting | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Javier Alberto Benchimol, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 1950
Record Dates: First submitted 2014-10-16; First posted 2014-10-31 (Estimated); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Hip Fracture
Keywords: hip fracture, elderly
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hip fracture: aged >65 with hip fracture

SUMMARY:
The purpose of this study is to create an institutional and population-based registry of Hip fracture in the elderly with a prospective survey based on epidemiological data, risk factors, diagnosis, prognosis, treatment, monitoring and survival.

DETAILED DESCRIPTION:
All patients over 65 years old who are admitted to the orthopedic and traumatology ward diagnosed with hip fracture will be assessed.

The generation of the list of potentially evaluable patients will be performed daily.

Once defined patient inclusion, an intern take oral informed consent and will proceed to complete the CRF.

Cohort will be followed at 3 months and a second follow-up at year.

Variables to be measured:

Patient Data Comorbidities Charlson score Scales functionality Factors prior to the fall Medications Trauma variables Complications Mortality

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 65 with hip fracture.
2. Admission to HIBA
3. Followed by any health care provider. -

Exclusion Criteria:

1 Patient refuses to participate in the registration or informed consent process

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: aged >65 hip fracture
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-11; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
mortality | 1 year

SECONDARY OUTCOMES:
frailty (measured by the Rockwood Scale) | 1 year
  It will performed once included in the Register the Rockwood Scale of Frailty and year follow-up after.

CONTACTS AND LOCATIONS:
Overall Officials: Javier A Benchimol, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolinsky FD, Fitzgerald JF, Stump TE. The effect of hip fracture on mortality, hospitalization, and functional status: a prospective study. Am J Public Health. 1997 Mar;87(3):398-403. doi: 10.2105/ajph.87.3.398. PMID 9096540
- [Background] Hannan EL, Magaziner J, Wang JJ, Eastwood EA, Silberzweig SB, Gilbert M, Morrison RS, McLaughlin MA, Orosz GM, Siu AL. Mortality and locomotion 6 months after hospitalization for hip fracture: risk factors and risk-adjusted hospital outcomes. JAMA. 2001 Jun 6;285(21):2736-42. doi: 10.1001/jama.285.21.2736. PMID 11386929
- [Background] Alarcon Alarcon T, Gonzalez-Montalvo JI. [Osteoporotic hip fracture. Predictive factors of short-and long-term functional recovery]. An Med Interna. 2004 Feb;21(2):87-96. doi: 10.4321/s0212-71992004000200010. No abstract available. Spanish. PMID 14974897
- [Background] Robinson TN, Eiseman B, Wallace JI, Church SD, McFann KK, Pfister SM, Sharp TJ, Moss M. Redefining geriatric preoperative assessment using frailty, disability and co-morbidity. Ann Surg. 2009 Sep;250(3):449-55. doi: 10.1097/SLA.0b013e3181b45598. PMID 19730176
- [Background] Riera-Espinoza G. Epidemiology of osteoporosis in Latin America 2008. Salud Publica Mex. 2009;51 Suppl 1:S52-5. doi: 10.1590/s0036-36342009000700009. PMID 19287895
- [Derived] Benchimol J, Fiorentini F, Elizondo CM, Boietti BR, Carabelli G, Barla J, Sancineto C, Waisman GD, Giunta DH. Institutional Registry of Elderly Patients With Hip Fracture in a Community-Based Tertiary Care Hospital in Argentina (RIAFC). Geriatr Orthop Surg Rehabil. 2016 Sep;7(3):121-5. doi: 10.1177/2151458516651309. Epub 2016 Jun 15. PMID 27551569

DOCUMENTS (1):
  • Study Protocol (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT02279550/Prot_000.pdf